CLINICAL TRIAL: NCT01573143
Title: Statin Therapy In Cardiac Surgery
Acronym: STICS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Chinese Academy of Medical Sciences (Other); Peking Union Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2.0 /06.09.11
Record Dates: First submitted 2012-02-13; First posted 2012-04-06 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Atrial Fibrillation; Myocardium; Injury
Keywords: Surgical Procedures, Cardiac; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Rosuvastatin; Post operative atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Wounds and Injuries | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Rosuvastatin (Experimental): Rosuvastatin (20 mg od)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin (20 mg od) started not earlier than 8 days before surgery and continued until the 5th post-operative day included;
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Placebo — Placebo started not earlier than 8 days before surgery and continued until the 5th post-operative day included.
  Arms: Sugar pill

SUMMARY:
The purpose of STICS trial (Statin Therapy In Cardiac Surgery) is to test whether perioperative treatment with Rosuvastatin 20 mg once daily prevents post-operative atrial fibrillation and reduces perioperative irreversible myocardial damage in patients undergoing elective cardiac surgery.

DETAILED DESCRIPTION:
Evidence that pre- or perioperative statin treatment may reduce the occurrence of post-operative atrial fibrillation and improve clinical outcome in patients undergoing coronary artery bypass graft (CABG) or major vascular surgery has been largely generated by observational studies. In a recent meta-analysis of 6 randomized trials (of which only 2 had postoperative atrial fibrillation (AF) as a predefined outcome) evaluating the use of perioperative statin treatment in patients undergoing cardiac surgery (n=651 patients in total - study size between 40 and 200 patients), statin use was found to reduce the patients' relative risk of developing postoperative AF by 43% (RR 0.57, 95%CI 0.45,0.72) and their absolute risk by 14% (95% CI 8%,20%). Although these findings would be consistent with a rapid and, possibly, lipid-independent antiarrhythmic effect of statins, they have important limitations (e.g., single-centre, small size, lack of continuous ECG monitoring, mostly "ancillary" findings") and less bearing on current clinical practice, as they mostly included statin-naïve patients. For these reasons, the recent guidelines for the management of AF have not given a strong recommendation for the use of statins in the prevention of postoperative AF. Thus, whether intensive statin treatment in the perioperative period is associated with prevention of AF, cardio protection, and improved clinical outcome remains to be demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients awaiting elective cardiac surgery who are willing and able to give informed consent for participation in the study and who are in sinus rhythm and not taking any antiarrhythmic medication, other than beta-adrenergic blocking agents, at the time of surgery.

Exclusion Criteria:

* History of obstructive hepato-biliary disease or other serious hepatic disease
* Untreated hypothyroidism
* Creatinine > 200 umol/L
* Personal and family history of hereditary muscle disorders
* Known intolerance to statins or history of muscle toxicity with fibrates or statins.
* On-going use of fibrates, niacin or of agents that are strong inhibitors of cytochrome P-450 or the P-glycoprotein within a month preceding randomization (cyclosporine, oral azole antifungals,macrolide antibiotics, protease inhibitors, nefazodone, amiodarone or ≥ 1L/day of grapefruit juice)
* Significant mitral valve disease (moderate or severe mitral regurgitation-eg. > grade II and/or mitral stenosis & mitral annular calcification).
* Patients treated with any anti-arrhythmic agent (other than beta-adrenergic receptor blockers).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1922 (Actual)
Dates: Start 2011-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Post operative atrial fibrillation detected on continuous ECG monitoring. | Monitoring will commence soon after surgery and will be continued until the end of post operative day 5
Myocardial injury assessed by Troponin release | Serial blood samples for Troponin assay will be collected at 6, 24, 48 and 120 hours after surgery

SECONDARY OUTCOMES:
Hospital and intensive care unit stay | Participants will be followed for the duration of the post operative period up to the day of initial discharge from the hospital, an expected average of 7 days.
Major in-hospital cardiac and/or cerebrovascular events (such as death, stroke, myocardial infarction,heart failure) and acute kidney injury | Participants will be followed for the duration of the post operative period up to the day of initial discharge from the hospital, an expected average of 7 days.
  Outcomes will be monitored for their presence/absence (Yes/No), the post operative day of event and duration as applicable.
Cardiac tissue and plasma/ urine biomarkers | Post operative period including day 5
  Cardiac tissue and plasma/ urine biomarkers of inflammation, oxidant stress, and cardiac function

CONTACTS AND LOCATIONS:
Overall Officials: Rory Collins, FRCP. FMed Sci, Study Chair — Clinical Trial Service Unit (CTSU), University of Oxford; Shenshou Hu, MD.PhD, Study Chair — Chinese Academy of Medical Sciences, Fuwai Hospital; Barbara Casadei, MD.DPhil.FRCP, Principal Investigator — Department of Cardiovascular Medicine, John Radcliffe Hospital, University of Oxford; Zheng Zhe, MD.PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Laufs U, Kilter H, Konkol C, Wassmann S, Bohm M, Nickenig G. Impact of HMG CoA reductase inhibition on small GTPases in the heart. Cardiovasc Res. 2002 Mar;53(4):911-20. doi: 10.1016/s0008-6363(01)00540-5. PMID 11922901
- [Background] Maack C, Kartes T, Kilter H, Schafers HJ, Nickenig G, Bohm M, Laufs U. Oxygen free radical release in human failing myocardium is associated with increased activity of rac1-GTPase and represents a target for statin treatment. Circulation. 2003 Sep 30;108(13):1567-74. doi: 10.1161/01.CIR.0000091084.46500.BB. Epub 2003 Sep 8. PMID 12963641
- [Background] Kim YM, Guzik TJ, Zhang YH, Zhang MH, Kattach H, Ratnatunga C, Pillai R, Channon KM, Casadei B. A myocardial Nox2 containing NAD(P)H oxidase contributes to oxidative stress in human atrial fibrillation. Circ Res. 2005 Sep 30;97(7):629-36. doi: 10.1161/01.RES.0000183735.09871.61. Epub 2005 Aug 25. PMID 16123335
- [Background] Kim YM, Kattach H, Ratnatunga C, Pillai R, Channon KM, Casadei B. Association of atrial nicotinamide adenine dinucleotide phosphate oxidase activity with the development of atrial fibrillation after cardiac surgery. J Am Coll Cardiol. 2008 Jan 1;51(1):68-74. doi: 10.1016/j.jacc.2007.07.085. PMID 18174039
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Chen WT, Krishnan GM, Sood N, Kluger J, Coleman CI. Effect of statins on atrial fibrillation after cardiac surgery: a duration- and dose-response meta-analysis. J Thorac Cardiovasc Surg. 2010 Aug;140(2):364-72. doi: 10.1016/j.jtcvs.2010.02.042. Epub 2010 Apr 9. PMID 20381820
- [Background] Reilly SN, Jayaram R, Nahar K, Antoniades C, Verheule S, Channon KM, Alp NJ, Schotten U, Casadei B. Atrial sources of reactive oxygen species vary with the duration and substrate of atrial fibrillation: implications for the antiarrhythmic effect of statins. Circulation. 2011 Sep 6;124(10):1107-17. doi: 10.1161/CIRCULATIONAHA.111.029223. Epub 2011 Aug 15. PMID 21844076
- [Background] Antoniades C, Bakogiannis C, Leeson P, Guzik TJ, Zhang MH, Tousoulis D, Antonopoulos AS, Demosthenous M, Marinou K, Hale A, Paschalis A, Psarros C, Triantafyllou C, Bendall J, Casadei B, Stefanadis C, Channon KM. Rapid, direct effects of statin treatment on arterial redox state and nitric oxide bioavailability in human atherosclerosis via tetrahydrobiopterin-mediated endothelial nitric oxide synthase coupling. Circulation. 2011 Jul 19;124(3):335-45. doi: 10.1161/CIRCULATIONAHA.110.985150. Epub 2011 Jul 5. PMID 21730307
- [Background] Antoniades C, Demosthenous M, Reilly S, Margaritis M, Zhang MH, Antonopoulos A, Marinou K, Nahar K, Jayaram R, Tousoulis D, Bakogiannis C, Sayeed R, Triantafyllou C, Koumallos N, Psarros C, Miliou A, Stefanadis C, Channon KM, Casadei B. Myocardial redox state predicts in-hospital clinical outcome after cardiac surgery effects of short-term pre-operative statin treatment. J Am Coll Cardiol. 2012 Jan 3;59(1):60-70. doi: 10.1016/j.jacc.2011.08.062. PMID 22192670
- [Derived] Zeng Z, Li F, Gai S, Chen R, Wang P, Wang J, Yang Y, Chen J, Zhang X, Wang X, Han Y, Lei C, Li X, Liu H, Zheng Z. The effect of clonal hematopoiesis on long-term outcomes in patients undergoing coronary artery bypass grafting. BMC Med. 2025 May 30;23(1):322. doi: 10.1186/s12916-025-04140-9. PMID 40442635
- [Derived] Liu H, Xu Z, Sun C, Chen Q, Bao N, Chen W, Zhou Z, Wang X, Zheng Z. Perioperative urinary thromboxane metabolites and outcome of coronary artery bypass grafting: a nested case-control study. BMJ Open. 2018 Aug 30;8(8):e021219. doi: 10.1136/bmjopen-2017-021219. PMID 30166295
- [Derived] Zheng Z, Jayaram R, Jiang L, Emberson J, Zhao Y, Li Q, Du J, Guarguagli S, Hill M, Chen Z, Collins R, Casadei B. Perioperative Rosuvastatin in Cardiac Surgery. N Engl J Med. 2016 May 5;374(18):1744-53. doi: 10.1056/NEJMoa1507750. PMID 27144849